CLINICAL TRIAL: NCT07307716
Title: Investigating the Impact of Cleaning Protocols on Oral Microbial Ecology and Early Dysbiosis Markers on Orthodontic Clear Aligner Patients: A Randomized Cross-over Clinical Study
Brief Title: Clear Aligner Cleaning: Brushing, Chlorhexidine, and BlueM Effects on Oral Microbial Ecology and Periodontal Indices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riyadh Elm University (Other)
Responsible Party: Principal Investigator, Faisal Ali Althobaiti, Principal Investigator, Riyadh Elm University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REU-ORTHO-ECOALIGN-XO-01
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Gingivitis; Dental Plaque
Keywords: Clear aligners; Chlorhexidine; BlueM; Oxygen-based cleanser; Mechanical toothbrushing; Supragingival plaque; Aligner biofilm; Fusobacterium nucleatum; Prevotella intermedia; MMP-8; Plaque index; Gingival index; Bleeding on probing; Randomized crossover
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Intervention Model Description: Three 1-month periods in randomized sequence (ABC/BCA/CAB) with 1-week washouts between the groups. A = mechanical toothbrushing (fluoride toothpaste), B = chlorhexidine mouthwash, C = oxygen-based cleanser (BlueM). Algners changed every 10 days; water-only while aligners are in
Who Masked: Outcomes Assessor
Masking Description: Culture enumeration from plaque and retrieved aligners will be processed under coded labels (P1-P3) by a single trained operator (FA) who is masked to protocol assignment. Microscopy and clinical assessments will be conducted unblinded after decoding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence ABC: Brushing then CHX Mouthwash then BlueM (Experimental): Participant completes three 1-month periods in order (A to B to C), each separated by a 1-week washout. A = Mechanical toothbrushing with fluoride toothpaste (control); B = Chlorhexidine (CHX) mouthwash; C = Oxygen-based cleanser (BlueM). Trays are changed every 10 days; aligners are worn 22 h/day; water-only while aligners are in.
  Interventions: Behavioral: Mechanical toothbrushing (fluoride toothpaste); Drug: Chlorhexidine mouthwash (0.2%); Other: Oxygen-based cleanser
- Sequence BCA: CHX Mouthwash then BlueM then Brushing (Experimental): Participant completes three 1-month periods in order (B to C to A), each separated by a 1-week washout. A = Mechanical toothbrushing with fluoride toothpaste (control); B = CHX mouthwash; C = Oxygen-based cleanser (BlueM). Trays are changed every 10 days; aligners are worn 22 h/day; water-only while aligners are in.
  Interventions: Behavioral: Mechanical toothbrushing (fluoride toothpaste); Drug: Chlorhexidine mouthwash (0.2%); Other: Oxygen-based cleanser
- Sequence CAB: BlueM then Brushing then CHX Mouthwash (Experimental): Participant completes three 1-month periods in order (C to A to B), each separated by a 1-week washout. A = Mechanical toothbrushing with fluoride toothpaste (control); B = CHX mouthwash; C = Oxygen-based cleanser (BlueM). Trays are changed every 10 days; aligners are worn 22 h/day; water-only while aligners are in.
  Interventions: Behavioral: Mechanical toothbrushing (fluoride toothpaste); Drug: Chlorhexidine mouthwash (0.2%); Other: Oxygen-based cleanser

INTERVENTIONS:
Behavioral: Mechanical toothbrushing (fluoride toothpaste) — Control oral-hygiene period using mechanical toothbrushing with a fluoride-containing toothpaste, per standardized study instructions, for the assigned 1-month period. No chlorhexidine or oxygen-based cleanser is used during this period; aligners are removed for oral-hygiene procedures per protocol.
  Other Names: Colgate Total
Drug: Chlorhexidine mouthwash (0.2%) — Chlorhexidine mouthwash used per standardized study instructions for the assigned 1-month period. No oxygen-based cleanser is used during this period; aligners are removed for mouthrinse use and oral-hygiene procedures per protocol. A 1-week washout without cleaning products separates periods.
  Other Names: CHX
Other: Oxygen-based cleanser — Oxygen-based cleanser (BlueM) used per standardized study instructions for the assigned 1-month period. No chlorhexidine is used during this period; aligners are removed for product use and oral-hygiene procedures per protocol. A 1-week washout without cleaning products separates periods.
  Other Names: BlueM

SUMMARY:
This randomized crossover study will assess how three aligner-cleaning methods affect early supragingival oral microbial ecology and periodontal health in adults using clear aligners. Each participant will complete three (1-month) periods in a randomized sequence with (1-week) washouts between periods:

1. Mechanical toothbrushing with fluoride toothpaste (control),
2. Chlorhexidine (CHX) mouthwash, and
3. an oxygen-based cleanser (BlueM).

Primary ecological outcomes focus on early dysbiosis indicators Fusobacterium nucleatum and Prevotella intermedia measured on retrieved aligner inner-surface biofilm and on supragingival plaque at the gingival margin. Secondary outcomes include periodontal indices (plaque index, gingival index, bleeding on probing) at index teeth and the host inflammatory marker MMP-8 in matrix-paired extracts (plaque and aligner).

Study visits occur at baseline and at the end of each 1-month period. Supragingival plaque is collected from the upper and lower first molars and central incisors; used aligners are swabbed immediately after removal. Participants are instructed to wear aligners about 22 hours/day, change trays every 10 days, remove aligners for meals and oral hygiene, and drink only water while aligners are in.

Laboratory procedures include blinded culture enumeration under coded labels (performed by a single trained operator, FA), confocal laser scanning microscopy, and RNA isolation with species-specific qRT-PCR; microscopy is conducted unblinded after decoding. The study will determine whether chlorhexidine or an oxygen-based cleanser produces more favorable early ecological changes and periodontal outcomes than mechanical brushing alone in clear aligner therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Undergoing or scheduled for treatment with clear aligners (CA).
* Presence of upper and lower first molars and central incisors.
* Periodontal health at baseline (no sites with PD ≥ 4 mm; no clinical attachment loss at index teeth; BI/PI within normal limits).
* No periodontal therapy within the previous 6 months.
* Able and willing to comply with study instructions and follow-up visits; signed informed consent.
* Sufficient remaining CA treatment (clinician-estimated): ≥ 14 weeks to safely cover three 1 month protocol periods plus washouts.

Minimum planned aligners remaining: ≥ 11 aligners (assuming 10 days/aligner) or equivalent continuous CA duration per treating orthodontist.

Exclusion Criteria:

* Patients requiring orthognathic surgery
* Uncontrolled systemic diseases (e.g., uncontrolled diabetes mellitus, autoimmune disease).
* Pregnancy or lactation.
* Use of systemic antibiotics and/or anti-inflammatory drugs within the last 3 months.
* Periodontal therapy within the last 6 months.
* Current tobacco use (smoking/smokeless) or vaping.
* Limited/express CA plans (e.g., ≤ 11 aligners or expected completion < 14 weeks).

Anticipated early completion of CA or major treatment changes (e.g., switch to fixed appliances) within the next ~4 months.

- Extensive caries, defective restorations, or prostheses affecting index teeth/sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Fusobacterium nucleatum CFU in supragingival plaque at the gingival margin (index teeth) | Baseline and end of each 1-month period (end of Period 1, Period 2, Period 3); 1-week washouts between periods.
  Anaerobic culture enumeration (CFU) of Fusobacterium nucleatum from supragingival plaque collected along the gingival margin of upper/lower first molars and central incisors using the standardized swab/microbrush protocol. Species confirmation per SOP. Culture processing blinded under coded labels (P1-P3) by FA. Metric: CFU per specimen (report also as log10 CFU if analyzed).
Fusobacterium nucleatum CFU on retrieved aligner inner-surface biofilm | Baseline and end of each 1-month period (end of Period 1, Period 2, Period 3); 1-week washouts between periods.
  Anaerobic culture enumeration (CFU) of Fusobacterium nucleatum from a standardized inner-surface swab of the used aligner (zones corresponding to gingival margins of index teeth). Species confirmation per laboratory SOP. Culture processing blinded under coded labels (P1-P3) by a single trained operator (FA). Metric: CFU per specimen (report also as log10 CFU if analyzed).

SECONDARY OUTCOMES:
Prevotella intermedia CFU on retrieved aligner inner-surface biofilm | Baseline and end of each 1-month period (end of Period 1, Period 2, Period 3); 1-week washouts between periods.
  Anaerobic culture enumeration (CFU) of Prevotella intermedia from a standardized inner-surface swab of the used aligner (zones corresponding to the gingival margins of the index teeth).
Prevotella intermedia CFU in supragingival plaque at the gingival margin (index teeth) | Baseline and end of each 1-month period (end of Period 1, Period 2, Period 3); 1-week washouts between periods.
  Anaerobic culture enumeration (CFU) of Prevotella intermedia from supragingival plaque collected along the gingival margin of upper/lower first molars and central incisors using the study's standardized swab/microbrush protocol.
MMP-8 concentration/activity in matrix-paired plaque and aligner extracts | Baseline and end of each 1-month period (end of Period 1, Period 2, Period 3); 1-week washouts between periods.
  MMP-8 measured from paired extracts obtained from supragingival plaque and retrieved aligner inner-surface biofilm collected from the same participant at each time point.
Plaque Index (PI) at index teeth | Baseline and end of each 1-month period (end of Period 1, Period 2, Period 3).
  Plaque Index recorded at the upper and lower first molars and central incisors; six sites per tooth.
Gingival Index (GI) at index teeth | Baseline and end of each 1-month period (end of Period 1, Period 2, Period 3).
  Gingival Index recorded at the upper and lower first molars and central incisors; six sites per tooth.
Bleeding on Probing (BoP) at index teeth | Baseline and end of each 1-month period (end of Period 1, Period 2, Period 3).
  BoP recorded at the upper and lower first molars and central incisors; six sites per tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Faisal A Althobaiti, BDS, Principal Investigator — Riyadh Elm University; Dr. Nancy M Ajwa, MSc, Study Director — Riyadh Elm University
Locations (1):
- Riyadh Elm University - Orthodontic Clinics, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) sharing will follow Riyadh Elm University IRB and SFDA requirements. A de-identified dataset (microbiological counts/abundances, MMP-8 values, periodontal indices, randomization order, and minimal demographics) may be shared after primary publication, subject to IRB approval and a data-use agreement

REFERENCES:
- [Background] Heller D, Helmerhorst EJ, Gower AC, Siqueira WL, Paster BJ, Oppenheim FG. Microbial Diversity in the Early In Vivo-Formed Dental Biofilm. Appl Environ Microbiol. 2016 Jan 8;82(6):1881-8. doi: 10.1128/AEM.03984-15. PMID 26746720
- [Background] Zhao R, Huang R, Long H, Li Y, Gao M, Lai W. The dynamics of the oral microbiome and oral health among patients receiving clear aligner orthodontic treatment. Oral Dis. 2020 Mar;26(2):473-483. doi: 10.1111/odi.13175. Epub 2020 Jan 8. PMID 31418980
- [Background] Miguel YD, Alcântara PR, Toyofuku ACMM, Shimizu RH. Periodontal monitoring in orthodontic treatment with orthodontic aligners: proof of concept. Rev Odontol UNESP. 2024;53:e20240016. doi:10.1590/1807-2577.01624